CLINICAL TRIAL: NCT00228449
Title: A Phase 2, Open-label, Multi-center, Sequential, Dose Finding Study of the Safety, Pharmacodynamics, and Pharmacokinetics of Peginesatide Administered Intravenously for the Maintenance Treatment of Anemia in Chronic Hemodialysis Patients
Brief Title: Peginesatide for Anemia in Chronic Hemodialysis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Affymax (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFX01-03
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: Anemia; Chronic Kidney Disease; Chronic Renal Failure
Keywords: anemia; chronic kidney disease; CKD; chronic renal failure; CRF; dialysis; erythropoietin; EPO; erythropoiesis stimulating agent; ESA; Hematide™; hemodialysis; hemoglobin; Hb; Hgb; Omontys; peginesatide; red blood cell; red blood cell production
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — peginesatide; hematide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Cohort 1 (Experimental): Conversion from epoetin alfa to peginesatide with a conversion factor (CF) of 0.033: peginesatide dose administered intravenously once every 4 weeks (Q4W) for a total of up to 6 doses. No transition period between epoetin treatment and start of peginesatide treatment.
  Interventions: Drug: peginesatide
- Cohort 2 (Experimental): Conversion from epoetin alfa to peginesatide with a CF of 0.041: peginesatide dose administered intravenously Q4W for a total of 6 doses. No transition period between epoetin treatment and start of peginesatide treatment.
  Interventions: Drug: peginesatide
- Cohort 3 (Experimental): Conversion from epoetin alfa to peginesatide with a CF of 0.050: peginesatide dose administered intravenously Q4W for a total of 6 doses. No transition period between epoetin treatment and start of peginesatide treatment.
  Interventions: Drug: peginesatide
- Cohorts 4 and 9 (Experimental): Conversion from epoetin alfa to peginesatide with a CF of 0.050: peginesatide dose administered intravenously Q4W for a total of 6 doses. With transition period between epoetin treatment and start of peginesatide treatment.
  Interventions: Drug: peginesatide
- Cohort 5 (Experimental): Conversion from epoetin alfa to peginesatide with a CF of 0.066: peginesatide dose administered intravenously Q4W for a total of 6 doses. With transition period between epoetin treatment and start of peginesatide treatment.
  Interventions: Drug: peginesatide
- Cohort 6 (Experimental): Conversion from epoetin alfa to peginesatide with tiered peginesatide starting doses of 0.05, 0.075, 0.1 or 0.15 mg/kg based on total weekly doses of epoetin alfa . Doses were administered intravenously Q4W for a total of 6 doses. With transition period between epoetin treatment and start of peginesatide treatment.
  Interventions: Drug: peginesatide
- Cohorts 7 and 8 (Experimental): Conversion from epoetin alfa to peginesatide with tiered peginesatide starting doses of 0.05, 0.075, 0.1 or 0.15 mg/kg based on total weekly doses of epoetin alfa dose. Doses were administered intravenously Q4W for a total of 6 doses. No transition period between epoetin treatment and start of peginesatide treatment.
  Interventions: Drug: peginesatide
- Cohorts 10 and 11 (Experimental): Conversion from epoetin alfa to peginesatide with fixed peginesatide starting doses of 4, 6, 12 or 16 mg based on total weekly doses of epoetin alfa. Doses were administered intravenously Q4W for a total of 6 doses. No transition period between epoetin treatment and start of peginesatide treatment.
  Interventions: Drug: peginesatide

INTERVENTIONS:
Drug: peginesatide
  Other Names: Omontys; Hematide; AF37702 Injection

SUMMARY:
The purpose of this study is to evaluate the safety, pharmacodynamics (PD), and pharmacokinetics (PK) of multiple intravenous doses of peginesatide in participants with chronic kidney disease (CKD) who are on hemodialysis.

DETAILED DESCRIPTION:
This was a Phase 2, multicenter, open-label, sequential, dose-finding trial designed with up to 12 treatment cohorts of 15 participants per cohort. Each participant received an intravenous dose of peginesatide administered once every 4 weeks (Q4W) for a total of 6 doses. Dosage regimens varied by cohort. Participants were followed for a minimum of 42 days after the last administration of peginesatide.

ELIGIBILITY:
Inclusion Criteria:

* Participant is informed of the investigational nature of this study and has given written, witnessed informed consent in accordance with institutional, local, and national guidelines;
* Males or females ≥ 18 years of age. Pre-menopausal females (with the exception of those who are surgically sterile) must have a negative pregnancy test at screening; those who are sexually active must practice a highly effective method of birth control for at least 4 weeks prior to study start, and must be willing to continue contraception until at least 4 weeks after the last dose of study drug. A highly effective method of birth control is defined as one that results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence (only acceptable if practiced as a life-style and not acceptable if one who is sexually active practices abstinence only for the duration of the study) or vasectomized partner;
* Clinically stable on hemodialysis for ≥6 months prior to study drug administration;
* Urea clearance/volume (Kt/V) ≥ 1.2 within the 4 weeks prior to study drug administration;
* Epoetin alfa maintenance therapy of ≥ 60 and ≤ 375 U/kg/wk continuously prescribed for 8 weeks prior to study drug administration. In the last 3 weeks prior to study drug administration, variation in prescribed total weekly dose must be ≤ 25% from the mean of the last three prescribed total weekly doses;
* Three mid- or end-of-week hemoglobin values of ≥ 10.0 and ≤ 12.5 g/dL in the 3 weeks prior to study drug administration with ≤ 1.2 g/dL difference between the three values;
* One serum ferritin level ≥ 100 micrograms per liter (μg/L) or one transferrin saturation ≥ 20% or one reticulocyte hemoglobin content (CHr) ≥ 29 picograms within 4 weeks prior to study drug administration;
* One serum folate level above the lower limit of normal during the 4 weeks prior to study drug administration;
* One vitamin B12 level above the lower limit of normal during the 4 weeks prior to study drug administration;
* Weight ≥ 45 kilograms (kg) within the 4 weeks prior to study drug administration;
* One white blood cell count ≥ 3.0 x 10^9/L within 4 weeks prior to study drug administration; and
* One platelet count ≥ 100 x 10^9/L and ≤ 500 x 10^9/L within 4 weeks prior to study drug administration.

Exclusion Criteria:

* Known intolerance to erythropoiesis stimulating agents;
* History of antibodies to erythropoiesis stimulating agents or history of pure red cell aplasia;
* Known intolerance to parenteral iron supplementation;
* Red blood cell transfusion within 12 weeks prior to study drug administration;
* Hemoglobinopathy (e.g., homozygous sickle-cell disease, thalassemia of all types, etc.);
* Known hemolysis;
* Chronic, uncontrolled, or symptomatic inflammatory disease (e.g., rheumatoid arthritis, systemic lupus erythematosus, etc.);
* C-reactive protein greater than 30 mg/L within the 4 weeks prior to study drug administration;
* Moderate or significant infection within 2 weeks prior to study drug administration;
* Known coagulation disorder based on clinical context and laboratory [activated partial thromboplastin time (aPTT) or international normalized ratio (INR)] results;
* Temporary (untunneled) dialysis access catheter;
* Uncontrolled or symptomatic secondary hyperparathyroidism;
* Poorly controlled hypertension within the 4 weeks prior to study drug administration, per the Investigator's clinical judgment (e.g., systolic ≥ 170 mm Hg or diastolic ≥ 100 mm Hg on repeat readings);
* Any history of multiple significant drug allergies;
* History of severe or unstable reactive airway disease within the previous 10 years;
* Epileptic seizure in the 6 months prior to screening;
* Chronic congestive heart failure (New York Heart Association Class IV);
* High likelihood of early withdrawal or interruption of the study (e.g., myocardial infarction, severe or unstable coronary artery disease, stroke, respiratory, autoimmune, neuropsychiatric, or neurological abnormalities, liver disease including active hepatitis B or C, active HIV disease, or any other clinically significant medical disease or conditions in the prior 6 months that may, in the Investigator's opinion, interfere with assessment or follow-up of the patient);
* Evidence of malignancy within the past 5 years (except non-melanoma skin cancer which is not an exclusion criterion);
* Life expectancy < 12 months;
* Anticipated elective surgery during the study period; and
* Previous exposure to any investigational agent within 6 weeks prior to administration of study drug or planned receipt during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2005-07; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Average weekly hemoglobin and hemoglobin change from baseline | Baseline to Week 27

SECONDARY OUTCOMES:
Percentage of participants with hemoglobin within 1.0 gram per deciliter (g/dL) above or below baseline | Baseline to Week 25
Percentage of participants who maintain hemoglobin within 9.5-13.0 g/dL | Baseline to Week 25
Percentage of participants who maintain hemoglobin within 11.0-13.0 g/dL | Baseline to Week 25

CONTACTS AND LOCATIONS:
Overall Officials: Affymax, Study Director — Affymax, Inc.
Locations (14):
- United States (14):
  - Research Facility, Birmingham, Alabama
  - Research Facility, Pine Bluff, Arkansas
  - Research Facility, Los Angeles, California
  - Research Facility, Mountain View, California
  - Research Facility, Lauderdale Lakes, Florida
  - Research Facility, Pembroke Pines, Florida
  - Research Facility, Shreveport, Louisiana
  - Research Facility, Detroit, Michigan
  - Research Facility, Minneapolis, Minnesota
  - Research Facility, New York, New York
  - Research Facility, Canton, Ohio
  - Research Facility, Nashville, Tennessee
  - Research Facility, San Antonio, Texas
  - Research Facility, Norfolk, Virginia

REFERENCES:
- [Derived] Besarab A, Zeig SN, Martin ER, Pergola PE, Whittier FC, Zabaneh RI, Schiller B, Mayo M, Francisco CA, Polu KR, Duliege AM. An open-label, sequential, dose-finding study of peginesatide for the maintenance treatment of anemia in chronic hemodialysis patients. BMC Nephrol. 2012 Aug 30;13:95. doi: 10.1186/1471-2369-13-95. PMID 22935486